CLINICAL TRIAL: NCT03132272
Title: Efficacy of Immunoadsorption for Treatment of Persons With Alzheimer Dementia and Agonistic Autoantibodies Against alpha1A-adrenoceptor (IMAD)
Brief Title: Immunoadsorption for Treatment of Alzheimer's Disease
Acronym: IMAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruiting, difficulties in finding eligible patients
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201503IMAD; CIV-16-02-014668 (Other: EUDAMED-No.)
Record Dates: First submitted 2016-11-16; First posted 2017-04-27 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer Dementia
Keywords: ADAsorb apheresis; Globaffin adsorber; Agonistic Autoantibodies; Immunoadsorption; Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunoadsorption with Globaffin for Alzheimer Dementia (Experimental): Immunoadsorption with Globaffin
  Interventions: Device: Immunoadsorption with Globaffin

INTERVENTIONS:
Device: Immunoadsorption with Globaffin — Immunoadsorption for treatment of persons with Alzheimer Dementia
  Other Names: agonistic autoantibodies; alpha1A-adrenoceptor; Globaffin adsorber columns; ADAsorb apheresis

SUMMARY:
Efficacy of immunoadsorption for treatment of persons with Alzheimer dementia and agonistic autoantibodies against alpha1A-adrenoceptor.

DETAILED DESCRIPTION:
The IMAD trial outlined aims to ascertain whether the positive effects of immunoadsorption (IA) on slowing down dementia progression, shown in a pilot trial, can be replicated in a slightly larger number of subjects and to comprehensively investigate the effects by a combination of brain and vessel imaging along with cognitive tests and further state-of-the-art cardiovascular, cerebrovascular and laboratory examinations. If the trial results underpin the hypothesis that IA effectively counteracts pathophysiological impairments and dementia-related cognitive decline, it may open up a new treatment approach against dementia, namely the reversal or avoidance of further vascular damage by the removal of agonistic autoantibodies (agAAB) in agAAB-positive persons.

The aim of this study is (beside of safety) to demonstrate the stop of the vascular remodeling and cognition decline by immunoadsorption, a therapeutic method which is well established in cardiology and nephrology.

ELIGIBILITY:
Inclusion Criteria:

* 55-85 years of age
* Diagnosis of Alzheimer's disease
* Presence of agAAB against alpha1-adrenoceptor
* Mini mental state examination (MMSE) score between 19 and 26
* Written informed consent given

Exclusion Criteria:

* Haemanalysis:

  * Presence of autoantibodies against the N-methyl-D-aspartate (NMDA) receptor
  * Defective blood coagulation at time of inclusion
  * Severe protein deficiency disorders
  * manifest Vitamin/Folic acid deficiency (substitution allowed)
* Active infectious disease, or signs of ongoing infection with C-reactive protein (CRP) >10mmol/L
* Impaired renal function (serum creatinine >220 μmol/L)
* Any disease requiring immunosuppressive drugs or therapeutic antibodies
* Non curative treated malignant disease or another life-threatening disease with poor prognosis (survival less than 2 years), except for basal-cell carcinoma
* Unstable angina pectoris, atrioventricular block (AV block) 2./3. degree or symptomatic sick sinus syndrome without implanted pacemaker, history of myocardial infarct, bypass or other revascularization measures, valvular heart defect (≥ 2. Degree)
* Severely reduced left ventricular systolic function (LVEF < 30%) and/or heart failure symptoms according to New York Heart Association (NYHA) class III/IV
* Clinical manifestation of arterial disease, vascular surgery: No Arteria Carotis Interna (ACI) Stenosis > 60%, peripheral artery occlusive disease (PAOD) > IIb, NASCET, no clinical manifest apparent stroke in anamnesis, MRI: no diffusion disorder, no expired territorial stroke
* Endocrine disorder excluding diabetes mellitus
* Severe hepatic damages (CHILD-Score < 4)
* Severe mental disorders (bipolar disorder, schizophrenia, depression) requiring treatment
* Alcohol or drug abuse
* Drug therapy against dementia since less than 3 months
* Psychopharmacological drug therapy since less than 3 months
* Dialysis requirement
* MRI contraindications (e.g. heart pacemaker)
* Legal tutelage
* Previous treatments with IA or immunoglobulin
* Inability to undergo the study procedure (IA on five consecutive days with subsequent Immunoglobulin G (IgG) substitution)
* treatment with angiotensin-converting-enzyme inhibitors (ACE inhibitors) during the IA (angiotensin receptor blockers (AT-blockers) possible)
* Participation in any other clinical/interventional study within less than 30 days prior to screening date

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow, estimated by Arterial Spin Labeling MRI | Measurement at 4 times over a 12 months period: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Measurement of cerebral blood flow and evaluation of changes between baseline and condition after intervention over a 12 months period

SECONDARY OUTCOMES:
Cognition (changes/improvement/impairment) | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Measurement by Alzheimer's Disease Assessment Scale (ADAS-cog)
Cognition (changes/improvement/impairment) | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Measurement by Mini Mental Status Examination-2 (MMSE)
Cognition (changes/improvement/impairment) | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Measurement by California Verbal Learning Test (CVLT)
Cognition (changes/improvement/impairment) | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Measurement by Benton Test
Vascular effects | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Left ventricular ejection fraction (LVEF)
Vascular effects | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Endothelial function: measurement by Endo-PAT
Vascular effects | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Arterial stiffness: measurement by Endo-PAT
Vascular effects | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Arterial stiffness: measurement by Mobil-O-Graph (pulse wave analysis)
Vascular effects | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Oxygen saturation: transcutaneous oxygen pressure examinations by PRÉCISE 8008, Medicap
Renal function | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Nephrosonography: position, size and surface of kidneys, echogenicity, presence and assessment of cysts and tumors, calcifications, nephroliths
Renal function | Measurement at 4 times: before IA (= baseline), 1 month after IA, 6 months after IA, 12 months after IA
  Estimated glomerular Filtration rate (eGFR) using Modification of Diet in Renal Disease (MDRD) formula
Laboratory parameters in liquor associated with Alzheimer's disease | Measurement at 2 times: before IA (= baseline) and 12 months after IA
  Measurement of beta-amyloid and tau species concentrations in liquor (optional; only if subjects gave informed consent in lumbar puncture)

OTHER OUTCOMES:
Serum analytics | 12 months
  analysis of agonistic autoantibodies against alpha1A adrenoceptor and measurement of different biomarkers, metabolites associated with Alzheimer's disease in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Dörr, Prof.Dr.med., Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No